CLINICAL TRIAL: NCT05836948
Title: An Open-label, Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of SHR-9839 for Injection in Patients With Advanced Solid Tumors
Brief Title: The Clinical Study of SHR-9839 for Injection in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-9839-I-101
Record Dates: First submitted 2023-04-19; First posted 2023-05-01 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-9839 (Experimental): three stages: dose escalation, dose expansion and efficacy expansion.
  Interventions: Drug: SHR-9839

INTERVENTIONS:
Drug: SHR-9839 — Weekly fixed dose injection of SHR-9839

SUMMARY:
This study is an open-label, phase I clinical trial of SHR-9839 in patients with advanced solid tumors. The whole study is divided into three stages: dose escalation, dose expansion and efficacy expansion.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically or cytologically confirmed unresectable locally advanced or metastatic solid tumors which is relapsed or refractory to standard treatment, or lack of standard treatment, or standard treatment is not applicable currently;
2. Have at least one measurable tumor lesion per RECIST v1.1;
3. ECOG performance status of 0-1;
4. Life expectancy ≥ 12 weeks;
5. Adequate bone marrow and organ function;
6. Subjects must voluntarily agree to participate in the trial and sign a written informed consent form.

Exclusion Criteria:

1. Patients with active central nervous system metastases or meningeal metastases;
2. Received anti-tumor treatment such as chemotherapy, biotherapy, targeted therapy, immunotherapy, radical radiotherapy, or other unlisted clinical research drugs or treatments within 4 weeks prior to the first use of the study drug;
3. History of serious cardiovascular and cerebrovascular diseases;
4. Subjects who received>30Gy of radiation therapy within 4 weeks before the first medication, and those who received ≤ 30Gy of palliative radiation therapy within 7 days before the first medication;
5. Adverse reactions of previous anti-tumor treatment have not recovered to Grade ≤ 1 per NCI-CTCAE v5.0.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2023-05-18 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) or maximum administered dose (MAD) | On the first day of each week,4 weeks is a treatment cycle
  Incidence and category of dose limiting toxicities (DLTs) during the first 4 week cycle of SHR-9839 treatment
Recommended Phase 2 dose (RP2D) | From Day 1 to 90 days after last dose
  RP2D will be determined on the basis of evaluation on MTD/MAD, PK, PD, efficacy data in dose escalation and dose expansion stages.
Incidence and severity of adverse events (AEs)/serious adverse events (SAEs) ([CTCAE] v5.0) | From Day 1 to 90 days after last dose
  Assess safety and tolerability of SHR-9839 by way of adverse events (CTCAE v5.0).

SECONDARY OUTCOMES:
PK parameter: Tmax of SHR-9839 | approximately 10 months
  Time to maximum concentration of SHR-9839
PK parameter: Cmax of SHR-9839 | approximately 10 months
  Maximum concentration of SHR-9839
PK parameter: AUC0-t of SHR-9839 | Approximately 10 months
  Area under the concentration-time curve from time 0 to the last measurable concentration time point of SHR-9839
PK parameter: AUC0-∞ of SHR-9839 | Approximately 10 months
  Area under the concentration-time curve from time 0 to infinity of SHR-9839
Immunogenicity of SHR-9839 | Approximately 12 months
  Anti-SHR-9839 antibody (ADA)
Overall response rate (ORR) | Approximately within 36 months
  Evaluated using RECIST 1.1
Duration of response (DoR) | Approximately within 36 months
  Evaluated using RECIST 1.1
Disease control rate (DCR) | Approximately within 36 months
  Evaluated using RECIST 1.1
Progression-free survival (PFS) | Approximately within 36 months
  Evaluated using RECIST 1.1

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Tumor Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided